CLINICAL TRIAL: NCT06395103
Title: LIGHTBEAM-U01 Substudy 01A: A Phase 1/2 Substudy to Evaluate the Safety and Efficacy of Zilovertamab Vedotin in Pediatric and Young Adult Participants With Hematologic Malignancies or Solid Tumors
Brief Title: Substudy 01A: Zilovertamab Vedotin in Pediatric and Young Adult Participants With Hematologic Malignancies or Solid Tumors (MK-9999-01A/LIGHTBEAM-U01)
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9999-01A; MK-9999-01A (Other: MSD); LIGHTBEAM-U01 (Other: MSD); 2023-507178-41-00 (Registry Identifier: EU CT); U1111-1295-3459 (Registry Identifier: UTN)
Record Dates: First submitted 2024-02-01; First posted 2024-05-01 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: B-cell Acute Lymphoblastic Leukemia; Diffuse Large B-cell Lymphoma; Burkitt Lymphoma; Neuroblastoma; Ewing Sarcoma
MeSH Terms: conditions — Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Neuroblastoma; Sarcoma, Ewing

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Zilovertamab vedotin (Experimental): Participants receive escalating doses of zilovertamab vedotin via intravenous (IV) infusion on Day 1 of each 21-day cycle (every 3 weeks).
  Interventions: Biological: Zilovertamab vedotin

INTERVENTIONS:
Biological: Zilovertamab vedotin — Administered via IV infusion
  Other Names: MK-2140; VLS-101

SUMMARY:
Substudy 01A is part of a platform study. The purpose of this study is to assess the efficacy and safety of zilovertamab vedotin in pediatric participants with relapsed or refractory B-cell acute lymphoblastic leukemia (B-ALL), diffuse large B-cell lymphoma (DLBCL)/Burkitt lymphoma, or neuroblastoma and in pediatric and young adult participants with Ewing sarcoma.

ELIGIBILITY:
The main inclusion and exclusion criteria include but are not limited to the following:

Inclusion Criteria:

* For hematological malignancies: Confirmed diagnosis of B-precursor B-ALL or DLBCL/Burkitt lymphoma according to World Health Organization (WHO) classification of neoplasms of the lymphoid tissues.
* For solid tumor malignancies: Histologically confirmed diagnosis of neuroblastoma or Ewing sarcoma.

Exclusion Criteria:

* History of solid organ transplant.
* Clinically significant (ie, active) cardiovascular disease.
* Known history of liver cirrhosis.
* Ongoing Grade >1 peripheral neuropathy.
* Demyelinating form of Charcot-Marie-Tooth disease.
* Diagnosed with Down syndrome.
* Ongoing graft-versus-host disease (GVHD) of any grade or receiving systemic GVHD treatment or prophylaxis.
* History of human immunodeficiency virus (HIV) infection.
* Contraindication or hypersensitivity to any of the study intervention components.
* Received prior radiotherapy within 4 weeks of start of study intervention. Participants must have recovered from all radiation-related toxicities.
* Ongoing, chronic corticosteroid therapy (exceeding 10 mg daily of prednisone equivalent). Prednisone equivalent dosing must have been stable for at least 4 weeks before Cycle 1 Day 1 (C1D1).
* Received a strong cytochrome P450 3A4 (CYP3A4) inhibitor within 7 days or a strong CYP3A4 inducer within 14 days before the start of study intervention or expected requirement for chronic use of a strong CYP3A4 inhibitor or inducer during the study intervention period and for 30 days after the last dose of study intervention
* Received prior systemic anticancer therapy including investigational agents within 4 weeks before the first dose of study intervention (except for prophylactic intrathecal chemotherapy and/or cytoreductive therapy with steroids/hydroxyurea.
* Received a live or live-attenuated vaccine within 30 days before the first dose of study intervention. Administration of killed vaccines is allowed.
* Has received an investigational agent or has used an investigational device within 4 weeks prior to study intervention administration.
* Known additional malignancy that is progressing or has required active treatment within the past 1 year.
* Active infection requiring systemic therapy.
* Known history of Hepatitis B or known active Hepatitis C virus infection.
* Participants who have not adequately recovered from major surgery or have ongoing surgical complications.

Ages: 6 Months to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-08-16 (Actual); Primary Completion 2029-03-31 (Estimated); Study Completion 2029-03-31 (Estimated)

PRIMARY OUTCOMES:
Part 1: Number of Participants from 1 to <18 years of Age Who Experience a Dose-Limiting Toxicity (DLT) | Up to 42 days
  Number of participants experiencing toxicities that are possibly, probably, or definitely related to study therapy; that meet pre-defined severity criteria; and result in a change in the given dose.
Part 1: Number of Participants from 1 to <18 years of Age Who Experience One or More Adverse Events (AEs) | Up to approximately 60 months
  An AE is defined as any untoward medical occurrence associated with the use of a drug in a participant, whether or not considered drug related. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product and does not imply any judgment about causality. The number of participants in Part 1 who experience at least 1 AE will be presented.
Part 1: Number of Participants from 1 to <18 years of Age Who Discontinue Study Treatment Due to AEs | Up to approximately 60 months
  An AE is defined as any untoward medical occurrence associated with the use of a drug in a participant, whether or not considered drug related. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product and does not imply any judgment about causality. The number of participants in Part 1 who discontinue study treatment due to an AE will be presented.
Part 1: Number of Participants from 1 to <18 years of Age Who Receive Dose Modification Due to AEs | Up to approximately 60 months
  An AE is defined as any untoward medical occurrence associated with the use of a drug in a participant, whether or not considered drug related. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product and does not imply any judgment about causality. The number of participants in Part 1 who receive a dose modification due to an AE will be presented.
Part 1 and Part 2: Objective Response (OR) for Participants with B-Cell Acute Lymphoblastic Leukemia (B-ALL) | Up to approximately 60 months
  OR for participants with B-ALL is defined as complete response (CR) or complete response with incomplete hematologic recovery (CRi) based on investigator's assessment per Ponte-di-Legno Consortium criteria. For Part 1 and Part 2, the OR for participants with B-ALL as assessed by investigator will be presented.
Part 1 and Part 2: OR for Participants with Diffuse Large B-Cell Lymphoma (DLBCL)/Burkitt Lymphoma, Neuroblastoma, and Ewing Sarcoma | Up to approximately 60 months
  OR for participants with DLBCL/Burkitt lymphoma, neuroblastoma, and Ewing sarcoma is defined as complete response (CR) or partial response (PR) based on investigator's assessment per International Pediatric Non-Hodgkin Lymphoma (IPNHL) Response Criteria for participants with DLBCL/Burkitt lymphoma, per International Neuroblastoma Response Criteria (INRC) for neuroblastoma, and per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 for Ewing sarcoma. For Part 1 and Part 2, the OR for participants with DLBCL/Burkitt lymphoma, neuroblastoma, and Ewing sarcoma as assessed by investigator will be presented.

SECONDARY OUTCOMES:
Part 1 and Part 2: Area Under the Curve (AUC) of Total Antibody | Predose on Day 1 of Cycles 1, 2, 3, 4, 5, 6 and every 4 cycles thereafter, and at end of infusion on Day 1 of Cycles 1 and 3. Each cycle is 21 days. (Up to approximately 60 months)
  Blood samples collected at designated time points will be used to determine the AUC of total antibody.
Part 1 and Part 2: Maximum Plasma Concentration (Cmax) of Total Antibody | Predose on Day 1 of Cycles 1, 2, 3, 4, 5, 6 and every 4 cycles thereafter, and at end of infusion on Day 1 of Cycles 1 and 3. Each cycle is 21 days. (Up to approximately 60 months)
  Blood samples collected at designated time points will be used to determine the Cmax of total antibody.
Part 1 and Part 2: Plasma Trough Concentration (Ctrough) of Total Antibody | Predose on Day 1 of Cycles 1, 2, 3, 4, 5, 6 and every 4 cycles thereafter, and at end of infusion on Day 1 of Cycles 1 and 3. Each cycle is 21 days. (Up to approximately 60 months)
  Blood samples collected at designated time points will be used to determine the Ctrough of total antibody.
Part 1 and Part 2: Apparent Terminal Half-life (t1/2) of Total Antibody | Predose on Day 1 of Cycles 1, 2, 3, 4, 5, 6 and every 4 cycles thereafter, and at end of infusion on Day 1 of Cycles 1 and 3. Each cycle is 21 days. (Up to approximately 60 months)
  Blood samples collected at designated time points will be used to determine the t1/2 of total antibody.
Part 1 and Part 2: AUC of Antibody-Drug Conjugate (ADC) | Predose on Day 1 of Cycles 1, 2, 3, 4, 5, 6 and every 4 cycles thereafter, and at end of infusion on Day 1 of Cycles 1 and 3. Each cycle is 21 days. (Up to approximately 60 months)
  Blood samples collected at designated time points will be used to determine the AUC of ADC.
Part 1 and Part 2: Cmax of Antibody-Drug Conjugate (ADC) | ose on Day 1 of Cycles 1, 2, 3, 4, 5, 6 and every 4 cycles thereafter, and at end of infusion on Day 1 of Cycles 1 and 3. Each cycle is 21 days. (Up to approximately 60 months)
  Blood samples collected at designated time points will be used to determine the Cmax of ADC.
Part 1 and Part 2: Ctrough of Antibody-Drug Conjugate (ADC) | Predose on Day 1 of Cycles 1, 2, 3, 4, 5, 6 and every 4 cycles thereafter, and at end of infusion on Day 1 of Cycles 1 and 3. Each cycle is 21 days. (Up to approximately 60 months)
  Blood samples collected at designated time points will be used to determine the Ctrough of ADC.
Part 1 and Part 2: t1/2 of Antibody-Drug Conjugate (ADC) | Predose on Day 1 of Cycles 1, 2, 3, 4, 5, 6 and every 4 cycles thereafter, and at end of infusion on Day 1 of Cycles 1 and 3. Each cycle is 21 days. (Up to approximately 60 months)
  Blood samples collected at designated time points will be used to determine the t1/2 of ADC.
Part 1 and Part 2: AUC of Monomethyl Auristatin E (MMAE) | Predose on Day 1 of Cycles 1, 2, 3, 4, 5, 6 and every 4 cycles thereafter, and at end of infusion on Day 1 of Cycles 1 and 3. Each cycle is 21 days. (Up to approximately 60 months)
  Blood samples collected at designated time points will be used to determine the AUC of MMAE.
Part 1 and Part 2: Cmax of Monomethyl Auristatin E (MMAE) | Predose on Day 1 of Cycles 1, 2, 3, 4, 5, 6 and every 4 cycles thereafter, and at end of infusion on Day 1 of Cycles 1 and 3. Each cycle is 21 days. (Up to approximately 60 months)
  Blood samples collected at designated time points will be used to determine the Cmax of MMAE.
Part 1 and Part 2: Ctrough of Monomethyl Auristatin E (MMAE) | Predose on Day 1 of Cycles 1, 2, 3, 4, 5, 6 and every 4 cycles thereafter, and at end of infusion on Day 1 of Cycles 1 and 3. Each cycle is 21 days. (Up to approximately 60 months)
  Blood samples collected at designated time points will be used to determine the Ctrough of MMAE.
Part 1 and Part 2: t1/2 of Monomethyl Auristatin E (MMAE) | Predose on Day 1 of Cycles 1, 2, 3, 4, 5, 6 and every 4 cycles thereafter, and at end of infusion on Day 1 of Cycles 1 and 3. Each cycle is 21 days. (Up to approximately 60 months)
  Blood samples collected at designated time points will be used to determine the t1/2 of MMAE.
Part 2: Number of Participants Who Experience One or More Adverse Events (AEs) | Up to approximately 60 months
  An AE is defined as any untoward medical occurrence associated with the use of a drug in a participant, whether or not considered drug related. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product and does not imply any judgment about causality. The number of participants in Part 2 who experience at least 1 AE will be presented.
Part 2: Number of Participants Who Discontinue Study Treatment Due to AEs | Up to approximately 60 months
  An AE is defined as any untoward medical occurrence associated with the use of a drug in a participant, whether or not considered drug related. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product and does not imply any judgment about causality. The number of participants in Part 2 who discontinue study treatment due to an AE will be presented.
Part 2: Number of Participants Who Receive Dose Modification Due to AEs | Up to approximately 60 months
  An AE is defined as any untoward medical occurrence associated with the use of a drug in a participant, whether or not considered drug related. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product and does not imply any judgment about causality. The number of participants in Part 2 who receive a dose modification due to an AE will be presented.
Part 1 and Part 2: Incidence of Antidrug Antibodies (ADAs) to Zilovertamab Vedotin | Predose on Day 1 of Cycles 1, 2, 3, 4, 5, 6 and every 4 cycles thereafter. Each cycle is 21 days. (Up to approximately 60 months)
  Blood samples collected at designated timepoints will be used to determine the ADA response to zilovertamab vedotin. The incidence of ADAs over time will be presented.
Part 1 and Part 2: Duration of Response (DOR) | Up to approximately 60 months
  DOR is defined as the time from the first documented evidence of CR/CRi for B-ALL or CR/PR for DLBCL/Burkitt lymphoma, Ewing sarcoma, and neuroblastoma until disease progression or death due to any cause, whichever occurs first. For participants under 1-year of age, the time from the first dose will start from the first dose a participant receives during Part 2.
Part 1 and Part 2: Percentage of Participants with DLBCL/Burkitt Lymphoma Who Receive Stem Cell Transplant (SCT) | Up to approximately 60 months
  The percentage of participants with DLBCL/Burkitt Lymphoma who go on to receive SCT will be presented.
Part 1 and Part 2: Percentage of Participants with B-ALL Who Receive SCT | Up to approximately 60 months
  The percentage of participants with B-ALL who go on to receive SCT will be presented.
Part 1 and Part 2: Percentage of Participants with B-ALL Who Receive Chimeric Antigen Receptor T (CAR-T) | Up to approximately 60 months
  The percentage of participants with B-ALL who go on to receive CAR-T will be presented.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (66):
- United States (16):
  - Children's Hospital Los Angeles ( Site 1006), Los Angeles, California
  - Children's Hospital Colorado-Center for Cancer and Blood Disorders ( Site 1016), Aurora, Colorado
  - Yale New Haven Hospital ( Site 1012), New Haven, Connecticut
  - Johns Hopkins All Children's Hospital ( Site 1025), St. Petersburg, Florida
  - University of Iowa-Holden Comprehensive Cancer Center ( Site 1017), Iowa City, Iowa
  - Dana-Farber Cancer Institute ( Site 1013), Boston, Massachusetts
  - Corewell Health ( Site 1001), Grand Rapids, Michigan
  - Children's Mercy Hospital ( Site 1024), Kansas City, Missouri
  - Rutgers Cancer Institute of New Jersey ( Site 1008), New Brunswick, New Jersey
  - New York Medical College ( Site 1023), Valhalla, New York
  - Sanford Fargo Medical Center-Roger Maris Cancer Center ( Site 1003), Fargo, North Dakota
  - Oregon Health and Science University ( Site 1004), Portland, Oregon
  - Children's Hospital of Philadelphia (CHOP) ( Site 1021), Philadelphia, Pennsylvania
  - Sanford Children's Hospital-Sanford Children's Specialty Clinic ( Site 1015), Sioux Falls, South Dakota
  - University of Texas MD Anderson Cancer Center ( Site 1007), Houston, Texas
  - Intermountain - Primary Children's Hospital ( Site 1014), Salt Lake City, Utah
- Australia (2):
  - Sydney Children's Hospital ( Site 1997), Randwick, New South Wales
  - Queensland Children's Hospital-Oncology & Haematology ( Site 1996), Brisbane, Queensland
- UZ Gent ( Site 1428), Ghent, Oost-Vlaanderen, Belgium
- Brazil (4):
  - Hospital Erasto Gaertner-CEPEP - Pesquisa Clínica ( Site 1268), Curitiba, Paraná
  - Hospital de Clinicas de Porto Alegre ( Site 1265), Porto Alegre, Rio Grande do Sul
  - Fundação Pio XII - Hospital de Câncer de Barretos ( Site 1264), Barretos, São Paulo
  - Fundação Faculdade Regional de Medicina de São José do Rio Preto-Centro Integrado de Pesquisa ( Site 1267), São José do Rio Preto, São Paulo
- McGill University Health Centre-Pediatric HematologyOncology ( Site 1223), Montreal, Quebec, Canada
- Chile (3):
  - Hospital Luis Calvo Mackenna ( Site 1879), Santiago, Region M. de Santiago
  - Hospital Carlos Van Buren ( Site 1880), Valparaíso, Región de Valparaíso
  - Hospital Clínico Regional Dr. Guillermo Grant Benavente ( Site 1881), Concepción, Región del Biobío
- Colombia (3):
  - Hospital Pablo Tobon Uribe ( Site 1923), Medellín, Antioquia
  - Clinica de la Costa S.A.S.-Clinical Research Oncology & Hematology -Pediatric ( Site 1924), Barranquilla, Atlántico
  - IMAT S.A.S ( Site 1921), Montería, Departamento de Córdoba
- Czechia (2):
  - Detska nemocnice FN Brno ( Site 1388), Brno, Brno-mesto
  - Fakultni nemocnice v Motole-Klinika detske hematologie a onkologie ( Site 1387), Prague, Praha 5
- Rigshospitalet-Department of paediatrics and adolescent medicine, Section of Paed haem-onc ( Site 1467), Copenhagen, Capital Region, Denmark
- France (5):
  - CHU de Bordeaux. Hopital Pellegrin ( Site 1105), Bordeaux, Aquitaine
  - CENTRE LEON BERARD-IHOPE (pediatrric oncology) ( Site 1100), Lyon, Auvergne-Rhône-Alpes
  - Centre Hospitalier Universitaire de Nantes - Hôpital Femme-Enfant-Adolescent Chu De Nantes ( Site 1104), Nantes, Pays de la Loire Region
  - Assistance Publique Hôpitaux de Marseille - Hôpital de la Timone ( Site 1102), Marseille, Provence-Alpes-Côte d'Azur Region
  - Gustave Roussy ( Site 1103), Villejuif, Île-de-France Region
- Germany (4):
  - Universitaetsklinikum Tuebingen ( Site 1142), Tübingen, Baden-Wurttemberg
  - Universitaetsklinikum Koeln. Klinik und Poliklinik ( Site 1145), Cologne, North Rhine-Westphalia
  - Universitätsklinikum Münster - Albert Schweitzer Campus-Pädiatrische Hämatologie und Onkologie ( Site 1141), Münster, North Rhine-Westphalia
  - Charité Campus Virchow-Klinikum-Klinik für Pädiatrie mit Schwerpunkt Hämatologie und Onkologie ( Site 1143), Berlin
- Aghia Sophia Children's Hospital-First Department of Pediatrics, National and Kapodistrian Universi ( Site 1797), Athens, Attica, Greece
- Semmelweis Egyetem ( Site 1838), Budapest, Hungary
- Israel (2):
  - Rambam Health Care Campus-Pediatric Hemato-Oncology ( Site 1674), Haifa
  - Sheba Medical Center ( Site 1675), Ramat Gan
- Italy (3):
  - Fondazione IRCCS Istituto Nazionale dei Tumori-Pediatric Oncology ( Site 1552), Milan, Lombardy
  - Ospedale Pediatrico Bambino Gesù IRCCS-Dipartimento di Onco-Ematologia e Terapia Cellulare e Genica ( Site 1553), Rome, Roma
  - Ospedale Infantile Regina Margherita-S.C. Oncoematologia Pediatrica ( Site 1551), Torino
- Prinses Maxima Centrum voor Kinderoncologie ( Site 1510), Utrecht, Netherlands
- Narodny ustav detskych chorob ( Site 1592), Bratislava, Bratislava Region, Slovakia
- South Korea (2):
  - Seoul National University Hospital-Pediatrics ( Site 1972), Seoul
  - Asan Medical Center-Pediatrics - Pedicatric Oncology ( Site 1973), Seoul
- Spain (3):
  - Hospital Sant Joan de Déu-Pediatric Oncology Department ( Site 1717), Esplugas de Llobregat, Barcelona
  - Hospital Infantil Universitario Niño Jesús-Servicio de Onco-Hematología Pediátrica ( Site 1715), Madrid, Madrid, Comunidad de
  - Hospital Universitari Vall d'Hebron-Servei de Hematologia i Oncologia Pediatrica ( Site 1716), Barcelona
- Sahlgrenska Universitetssjukhuset ( Site 1634), Gothenburg, Västra Götaland County, Sweden
- National Taiwan University Hospital ( Site 1983), Taipei, Taiwan
- Turkey (Türkiye) (3):
  - Ege Universitesi Hastanesi ( Site 1963), Bornova, İzmir
  - Hacettepe Universite Hastaneleri ( Site 1961), Ankara
  - Ankara Bilkent Şehir Hastanesi ( Site 1962), Ankara
- United Kingdom (5):
  - Birmingham Children's Hospital-Oncology/Haematology ( Site 1349), Birmingham, England
  - Royal Victoria Infirmary-Great North Children's Hospital ( Site 1348), Newcastle upon Tyne, England
  - University College London Hospital ( Site 1350), London, London, City of
  - Royal Marsden Hospital (Sutton)-Drug Development Unit ( Site 1347), Sutton, Surrey
  - University Hospital of Wales ( Site 1346), Cardiff

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26269&tenant=MT_MSD_9011